CLINICAL TRIAL: NCT00694577
Title: Partial Breast Irradiation (PBI) for Selected Patients With Early Invasive or Non-Invasive Breast Cancer: A Phase I Feasibility/Pilot Study
Brief Title: Partial Breast Irradiation (PBI) for Selected Patients With Early Invasive or Non-Invasive Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Alphonse Taghian, MD, PhD, Professor of Radiation Oncology, Harvard Medical School, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 03-179
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Results first posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-10

CONDITIONS: Ductal Breast Cancer
Keywords: non-invasive breast cancer; early invasive breast cancer; radiation; PBI
MeSH Terms: conditions — Carcinoma, Ductal, Breast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Irradiation using 32 Gy / 8 fractions (Experimental): Study Participants 1-100 Partial Breast Irradiation using 32 Gy / 8 fractions BID in one week
  Interventions: Radiation: Partial Breast Irradiation using 32 Gy / 8 fractions; Radiation: Partial Breast Irradiation using 36 Gy / 9 fractions; Radiation: Partial Breast Irradiation using 40 Gy /10 fractions
- Irradiation using 36 Gy / 9 fractions (Experimental): Study Participants 101-200 Partial Breast Irradiation using 36 Gy / 9 fractions BID in one week
  Interventions: Radiation: Partial Breast Irradiation using 32 Gy / 8 fractions; Radiation: Partial Breast Irradiation using 36 Gy / 9 fractions; Radiation: Partial Breast Irradiation using 40 Gy /10 fractions
- Irradiation using 40 Gy / 10 fractions (Experimental): Study Participants 201-330 Partial Breast Irradiation using 40 Gy / 10 fractions BID in one week
  Interventions: Radiation: Partial Breast Irradiation using 32 Gy / 8 fractions; Radiation: Partial Breast Irradiation using 36 Gy / 9 fractions; Radiation: Partial Breast Irradiation using 40 Gy /10 fractions

INTERVENTIONS:
Radiation: Partial Breast Irradiation using 32 Gy / 8 fractions — 32 Gy-8 Treatments, 4 Treatment Days
  Other Names: PBI
Radiation: Partial Breast Irradiation using 36 Gy / 9 fractions — 36 Gy- 9 Treatments, 4 1/2 Treatment Days
  Other Names: PBI
Radiation: Partial Breast Irradiation using 40 Gy /10 fractions — 40 Gy-10 Treatments, 5 Treatment days
  Other Names: PBI

SUMMARY:
The purpose of this study is to determine the feasibility of partial breast irradiation in participants with early invasive or non-invasive breast cancer.

DETAILED DESCRIPTION:
* In this study, radiotherapy is given only to a portion of the breast around the tumor bed using external radiation treatments. This approach is called "partial breast irradiation".
* Participants will undergo a planning session for the radiation treatments. This planning will be done by CT scan days or weeks before the start of treatment. This planning process is the same as that used to plan conventional radiation therapy treatments.
* Radiation therapy will begin 4-12 weeks after the last surgery of the breast in individuals not receiving chemotherapy first. For individuals receiving chemotherapy before radiation therapy, radiation therapy will start 2-6 weeks after ending chemotherapy.
* We will be studying three levels of radiation doses to see which is best. The dose the participant receives will depend upon when they are enrolled on the trial.
* Participants will receive radiation treatment twice each day for 4 or 5 treatment days, with an overall treatment time of one week.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unicentric Stage I Invasive Ductal breast cancer. Histologically negative tumor margin 2mm or more from any inked edges, or no tumor in re-excision specimen or final shaved specimen.
* Patient may have been treated with adjuvant chemotherapy, or be on adjuvant hormonal therapy or begin hormonal therapy following XRT
* 18 years of age or older
* ECOG Performance Status 0
* Required laboratory data as outlined in the protocol

Exclusion Criteria:

* Multicentric IDC of the breast defined as discontiguous tumors separated by at least 5cm of uninvolved tissue
* Multifocal IDC of the breast, defined as discontiguous discrete foci of invasive carcinoma, separated by uninvolved intervening tissue, but within an overall span of 5cm, or within the same breast quadrant or subareolar central region
* Tumor > 2.0cm, nodal involvement, or metastatic involvement
* Histological evidence of: lymphovascular invasion; blood vessel invasion; extensive intraductal component; invasive lobular carcinoma and infiltrating carcinoma of mixed ductal and lobular type; DCIS with microinvasion and DCIS suspicious for microinvasion; infiltrating micropapillary carcinoma
* Known mutation carrier, including BRCA1 and BRCA2
* History of cosmetic or reconstructive breast surgery
* Psychiatric illness which would prevent the patient from giving informed consent
* Medical conditions such as uncontrolled infection, uncontrolled diabetes mellitus or connective tissue disease
* Participants with a "currently active" second malignancy other than non-melanoma skin cancers
* Patients with diffuse (> 1 quadrant or >5cm) suspicious microcalcifications
* Women who are pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2003-09; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse Taghian, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pashtan IM, Recht A, Ancukiewicz M, Brachtel E, Abi-Raad RF, D'Alessandro HA, Levy A, Wo JY, Hirsch AE, Kachnic LA, Goldberg S, Specht M, Gadd M, Smith BL, Powell SN, Taghian AG. External beam accelerated partial-breast irradiation using 32 gy in 8 twice-daily fractions: 5-year results of a prospective study. Int J Radiat Oncol Biol Phys. 2012 Nov 1;84(3):e271-7. doi: 10.1016/j.ijrobp.2012.04.019. Epub 2012 May 30. PMID 22652104
- [Derived] Recht A, Ancukiewicz M, Alm El-Din MA, Lu XQ, Martin C, Berman SM, Hirsch AE, Kachnic LA, Katz A, MacDonald S, Nedea EA, Stevenson MA, Powell SN, Taghian AG. Lung dose-volume parameters and the risk of pneumonitis for patients treated with accelerated partial-breast irradiation using three-dimensional conformal radiotherapy. J Clin Oncol. 2009 Aug 20;27(24):3887-93. doi: 10.1200/JCO.2008.20.0121. Epub 2009 Jul 20. PMID 19620489

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Irradiation Using 32 Gy / 8 Fractions | Irradiation Using 36 Gy / 9 Fractions | Irradiation Using 40 Gy / 10 Fractions
Started | 99 | 101 | 124
Completed | 98 | 101 | 124
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Study Participants 1-100
  Partial Breast Irradiation using 32 Gy / 8 fractions, BID: 4 Treatment Days, within 1 week
- Group 2: Study Participants 101-200
  Partial Breast Irradiation using 36 Gy / 9 fractions, BID: 4 1/2 Treatment Days, within 1 week
- Group 3: Study Participants 201-330
  Partial Breast Irradiation using 40 Gy / 10 fractions, BID: 5 Treatment Days, within 1 week
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 98 | 101 | 124 | 323
Age, Continuous [Median (Full Range); unit: years] | 61 [40 to 80] | 61 [40 to 87] | 60 [42 to 86] | 61 [40 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 101 | 124 | 323
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 98 | 101 | 124 | 323
Number of patients with triple negative cancer (ER-/PR-/HER2-) [Count of Participants; unit: Participants] — Number of patients with ER-/PR-/HER2- cancer.
  Participants | 10 | 4 | 2 | 16

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Local Control of Early Breast Cancer Treated by Partial Breast Irradiation Using Different Radiation Doses Determined by Completion.
Description: Feasibility and local control of early breast cancer treated by partial breast irradiation using different radiation doses. Number of patients who completed partial breast irradiation was used to determine feasibility.
Time Frame: 10 years
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Study Participants 1-100 Partial Breast Irradiation using 32 Gy / 8 fractions BID in one week
  Partial Breast Irradiation using 32 Gy / 8 fractions: 32 Gy-8 Treatments, 4 Treatment Days
  Partial Breast Irradiation using 36 Gy / 9 fractions: 36 Gy- 9 Treatments, 4 1/2 Treatment Days
  Partial Breast Irradiation using 40 Gy /10 fractions: 40 Gy-10 Treatments, 5 Treatment days
- Group 2: Study Participants 101-200 Partial Breast Irradiation using 36 Gy / 9 fractions BID in one week
  Partial Breast Irradiation using 32 Gy / 8 fractions: 32 Gy-8 Treatments, 4 Treatment Days
  Partial Breast Irradiation using 36 Gy / 9 fractions: 36 Gy- 9 Treatments, 4 1/2 Treatment Days
  Partial Breast Irradiation using 40 Gy /10 fractions: 40 Gy-10 Treatments, 5 Treatment days
- Group 3: Study Participants 201-330 Partial Breast Irradiation using 40 Gy / 10 fractions BID in one week
  Partial Breast Irradiation using 32 Gy / 8 fractions: 32 Gy-8 Treatments, 4 Treatment Days
  Partial Breast Irradiation using 36 Gy / 9 fractions: 36 Gy- 9 Treatments, 4 1/2 Treatment Days
  Partial Breast Irradiation using 40 Gy /10 fractions: 40 Gy-10 Treatments, 5 Treatment days
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 98 | 101 | 124
Participants | 98 | 101 | 124

2. Primary Outcome: Number of Patients Who Presented With Local Recurrence in the Same Breast Which Received Treatment and Confirmed by Positive Biopsy
Description: Risk of local failure after PBI determined by number of patients who presented with local recurrence in the same breast confirmed by positive biopsy
Time Frame: 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 98 | 101 | 124
Participants | 6 | 4 | 1

3. Secondary Outcome: Number of Patients Who Presented With Moderate to Severe Composite Toxicity as an Endpoint
Description: Number of patients who presented with moderate to severe composite toxicity as an endpoint
Time Frame: 8 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 98 | 101 | 124
Participants | 46 | 67 | 100

4. Secondary Outcome: Number of Patients Who Developed Moderate to Severe Breast Fibrosis After Partial Breast Irradiation
Description: Rate of moderate to severe breast fibrosis determined by number of patients who developed moderate to severe breast fibrosis after partial breast irradiation according to radiation dose level
Time Frame: 8 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 98 | 101 | 124
Participants | 37 | 52 | 83

5. Secondary Outcome: Number of Patients Who Had Poor/Fair Cosmetic Outcome After Partial Breast Irradiation
Description: Number of patients who had poor/fair cosmetic outcome after partial breast irradiation. Other participants had excellent/good cosmetic outcomes.
Time Frame: 8 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 98 | 101 | 124
Participants | 21 | 36 | 56

6. Secondary Outcome: To Evaluate Patient Satisfaction
Description: A survey asking the patient about her level of satisfaction with her PBI treatment. Patients who are totally satisfied with their appearance.
Time Frame: 8 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 98 | 101 | 124
Participants | 94 | 94 | 110

ADVERSE EVENTS:
Time Frame: 8 years
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/99 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/99 | 0/124
Other Adverse Events (participants affected / at risk) | 0/98 | 0/99 | 0/124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-04-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT00694577/Prot_SAP_000.pdf
  • Informed Consent Form (2009-10-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT00694577/ICF_001.pdf